CLINICAL TRIAL: NCT07189481
Title: Evaluation Einer Team Time-out Checkliste im OP
Brief Title: Design and Evaluation of a Team Timeout Checklist (TTOC) to Improve Information Exchange in the Operating Room Before Skin Incision
Acronym: TTOC
Status: Completed | Type: Observational
Sponsor: University of Jena (Other)
Collaborators: University of Leipzig (Other)
Responsible Party: Principal Investigator, Mona Weiss, Professor Mona Weiss, PhD, University of Jena
Other Study IDs: University of Leipzig Ethics
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2024-06

CONDITIONS: Checklist; Teamwork; Information Exchange
Keywords: checklist; timeout; teamwork; communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pre-post intervention study: teams were observed before and after checklist use

SUMMARY:
In this study, we designed and evaluated a team timeout checklist (TTOC) which aimed at improving team communication and information exchange before skin incision. The WHO surgical safety checklist was used as a basis with the following changes: we clarified the wording of specific items (e.g., surgical site), we clarified checks by denoting separate items involved for each check, and we denoted circulating nurses as responsible for checklist readout and adherence.

ELIGIBILITY:
Inclusion Criteria: Personnel working in the operating room (nurses, surgeons, anesthesiologists, technical support staff)

-

Exclusion Criteria:

* anyone who did not give their oral consent to be observed during surgeries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OR personnel working in orthopedics and traumatology: surgeons, anesthesiologists, anesthesia nurses, circulating nurses, technical support staff
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
information exchange | from the time patients were rolled into the OR until skin incision
  this measure assessed whether all sub-items on the TTOC were adequately checked and respective information audibly shared in the team
team communication | from the time patients were rolled into the OR until skin incision
  using a validate coding scheme, we assessed how team members communicated with each other using professional coding software to log a set of ten behaviors (e.g., instructions, questions, confirmations, speaking up...)

SECONDARY OUTCOMES:
duration of pre skin incision period with and without checklist | from the time patients were rolled into the OR until skin incision
  to assess how long the period before incision takes with and without TTOC

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leipzig, Leipzig, Germany